CLINICAL TRIAL: NCT01848522
Title: Creation and Setting up of Therapeutic Programs, Interprofessional Communication, Patients' Education and Counseling: a Qualitative Study in 3 Physical Therapy and Rehabilitation Departments
Brief Title: Creation and Setting up of Therapeutic Programs, Interprofessional Communication, Patients' Education and Counseling
Acronym: EMCIQUAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10043
Record Dates: First submitted 2013-04-30; First posted 2013-05-07 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Professionals and Patients in the Department of Physical Medicine and Rehabilitation
Keywords: qualitative study; rehabilitation; physical therapy; patient education; health care; administration; patient satisfaction; handicap
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to suggest system for improving patients' management through a detail analysis of physical therapy departments functioning

DETAILED DESCRIPTION:
First phase:

* Description of the actual patients' management through individual semi directive interviews and focus groups of health professionals, patients, and members of the hospital directory departments.
* Identification of barriers

Second phase: suggestion of system for improving patients' management

ELIGIBILITY:
Inclusion Criteria:

* For doctors: affiliation to physical therapy and rehabilitation departments, age, career and function
* For other health professionals: affiliation to physical therapy and rehabilitation departments, service length, age, gender
* For patients: age, gender and therapeutic programs

Exclusion Criteria:

- Persons not wishing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each of 3 centers, we will evaluate :
  * 13 healthcare professionals
  * 8 patients
  * 1 hospital executives
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Patient management system | 1 year
  Qualitative study in the form of semi-structured individual interviews and group meetings (focus group) with health professionals, patients (and members of the hospital management to collect comprehensive information, prior to the formalization and implementation of specific actions.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Poiraudeau, MD, PhD, Principal Investigator — AP-HP, Descartes University, INSERM
Locations (3):
- France (3):
  - CHU Henri Mondor-Albert Chenevier, Créteil
  - CHU Raymond Poincaré- Groupement hospitalier universitaire Ouest, Garches
  - Cochin Hospital, Paris

REFERENCES:
- [Background] Coudeyre E, Rannou F, Tubach F, Baron G, Coriat F, Brin S, Revel M, Poiraudeau S. General practitioners' fear-avoidance beliefs influence their management of patients with low back pain. Pain. 2006 Oct;124(3):330-337. doi: 10.1016/j.pain.2006.05.003. Epub 2006 Jun 5. PMID 16750297
- [Background] Coudeyre E, Tubach F, Rannou F, Baron G, Coriat F, Brin S, Revel M, Poiraudeau S. Effect of a simple information booklet on pain persistence after an acute episode of low back pain: a non-randomized trial in a primary care setting. PLoS One. 2007 Aug 8;2(8):e706. doi: 10.1371/journal.pone.0000706. PMID 17684553
- [Background] Poiraudeau S, Rannou F, Le Henanff A, Coudeyre E, Rozenberg S, Huas D, Martineau C, Jolivet-Landreau I, Revel M, Ravaud P. Outcome of subacute low back pain: influence of patients' and rheumatologists' characteristics. Rheumatology (Oxford). 2006 Jun;45(6):718-23. doi: 10.1093/rheumatology/kei231. Epub 2005 Dec 23. PMID 16377729
- [Background] Ravaud P, Flipo RM, Boutron I, Roy C, Mahmoudi A, Giraudeau B, Pham T. ARTIST (osteoarthritis intervention standardized) study of standardised consultation versus usual care for patients with osteoarthritis of the knee in primary care in France: pragmatic randomised controlled trial. BMJ. 2009 Feb 23;338:b421. doi: 10.1136/bmj.b421. PMID 19237406
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Coudeyre E, Demaille-Wlodyka S, Poizat S, Burton K, Hamonet MA, Revel M, Poiraudeau S. Could a simple educational intervention modify beliefs about whiplash? A preliminary study among professionals working in a rehabilitation ward. Ann Readapt Med Phys. 2007 Oct;50(7):552-7, 545-51. doi: 10.1016/j.annrmp.2007.05.005. Epub 2007 Jun 18. English, French. PMID 17597246
- [Background] Coudeyre E, Givron P, Vanbiervliet W, Benaim C, Herisson C, Pelissier J, Poiraudeau S. [The role of an information booklet or oral information about back pain in reducing disability and fear-avoidance beliefs among patients with subacute and chronic low back pain. A randomized controlled trial in a rehabilitation unit]. Ann Readapt Med Phys. 2006 Nov;49(8):600-8. doi: 10.1016/j.annrmp.2006.05.003. Epub 2006 May 26. French. PMID 16793163